CLINICAL TRIAL: NCT01351675
Title: Bardoxolone Methyl Evaluation in Patients With Chronic Kidney Disease and Type 2 Diabetes: the Occurrence of Renal Events (BEACON)
Brief Title: Bardoxolone Methyl Evaluation in Patients With Chronic Kidney Disease and Type 2 Diabetes
Acronym: BEACON
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IDMC recommendation for safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-0903
Record Dates: First submitted 2010-12-03; First posted 2011-05-11 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2
Keywords: Chronic kidney disease; Type 2 diabetes; Diabetic nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Bardoxolone Methyl (Experimental)
  Interventions: Drug: Bardoxolone Methyl: 20 mg

INTERVENTIONS:
Drug: Placebo — Oral, once daily
  Arms: Placebo
Drug: Bardoxolone Methyl: 20 mg — 20 mg, oral, once daily
  Other Names: RTA-402
  Arms: Bardoxolone Methyl

SUMMARY:
This study assesses the efficacy of bardoxolone methyl relative to placebo in delaying progression to end-stage renal disease (ESRD) and cardiovascular deaths in patients with Stage 4 Chronic Kidney Disease (CKD) and type 2 diabetes receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Screening eGFR ≥ 15.0 and < 30.0 mL/min/1.73 m2;
2. A history of type 2 diabetes; diagnosis should have been made at ≥ 30 years of age;
3. Male or female at least 18 years of age;
4. Treatment with an angiotensin converting enzyme (ACE)inhibitor and/or an angiotensin II receptor blocker (ARB)for at least 6 weeks prior to and during screening. Stable dose 2 weeks prior to and during screening. Patients not taking an ACE inhibitor and/or ARB because of a medical contraindication must have discontinued treatment at least 8 weeks prior to Screening Visit A;
5. Mean systolic blood pressure (SBP) must be ≤ 160 mmHg and ≥ 105 mmHg and mean diastolic blood pressure (DBP) must be < 90 mm Hg during screening; both mean SBP and mean DBP (determined as the average of three readings) must be within this range at two separate time points measured at least 4 days apart during the screening period (blood pressure may be re-evaluated once during an unscheduled visit);
6. Willing to practice methods of birth control (both male and female patients) during the entire study period and for at least 30 days after the last dose of the study drug is ingested;
7. Serum magnesium level must be ≥ 1.3 mEq/L (0.65 mmol/L) at Screening Visit B or during subsequent unscheduled visit during screening (serum magnesium level may be re-evaluated once during an unscheduled visit);
8. Willing and able to cooperate with all aspects of the protocol;
9. Willing and able to give written informed consent for study participation and provide consent for access to medical data according to appropriate local data protection legislation, allowing authorization to access medical records and describe events captured in the endpoints

Exclusion Criteria:

1. Type 1 diabetes mellitus (juvenile onset). If a history of diabetic ketoacidosis exists, a C-peptide level must confirm type 2 diabetes;
2. Known non-diabetic renal disease (e.g., polycystic kidney disease, focal segmental glomerulosclerosis) [nephrosclerosis superimposed on diabetic kidney disease is acceptable];
3. Ongoing clinical evidence suggesting non-diabetic renal disease other than nephrosclerosis;
4. History of a renal transplant or a planned transplant from a living donor during the study;
5. Albumin to creatinine ratio (ACR) greater than 3500 mg/g (395.5 mg/mmol);
6. Hemoglobin A1c level > 11.0% (97 mmol/mol) during screening;
7. Acute dialysis or acute kidney injury within 12 weeks prior to screening or during screening;
8. Clinical signs and/or symptoms of uremia and expected need for renal replacement therapy within 12 weeks following randomization, as assessed by the investigator;
9. Recently active cardiovascular disease defined as: a. Unstable angina pectoris within 12 weeks before study randomization; b. Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 12 weeks before study randomization; c. Cerebrovascular accident, including transient ischemic attack within 12 weeks before study randomization; d. Current diagnosis of Class III or IV New York Heart Association (NYHA) congestive heart failure;
10. Clinical diagnosis of severe obstructive valvular heart disease or severe obstructive hypertrophic cardiomyopathy;
11. Atrioventricular block, 2o or 3o, not successfully treated with a pacemaker;
12. DAdministration of a contrast agent that may induce nephropathy within 30 days prior to study randomization or planned during the study;
13. Systemic immunosuppression for a total of > 2 weeks, cumulatively, within the 12 weeks prior to randomization or planned during the study;
14. Total bilirubin, aspartate aminotransaminase (AST) or alanine aminotransaminase (ALT) levels greater than the upper limit of normal (ULN), or alkaline phosphatase level greater than two times the ULN on ANY screening laboratory test result;
15. Female patients who are pregnant, intend to become pregnant during the study, or are nursing;
16. BMI < 18.5 g/m2
17. Known hypersensitivity to any component of the study drug;
18. Current history of drug or alcohol abuse as assessed by the investigator;
19. Clinically significant infection requiring intravenous administration of antibiotics or hospitalization within 6 weeks of screening or during screening;
20. Hepatitis B surface antigen positive;
21. Diagnosis or treatment of a malignancy in the past 5 years, excluding non-melanoma skin cancer and carcinoma in situ of the cervix or a condition highly likely to transform into malignancy during the course of the study;
22. A clinical condition that in the judgment of the investigator could potentially pose a health risk to the patient while involved in the study;
23. Participation in a clinical study involving any intervention within 30 days prior to randomization, concurrent participation in such a study, or participation in a prior clinical study involving bardoxolone methyl in any form;
24. Unable to communicate or cooperate with the investigator due to language problems, poor mental development or impaired cerebral function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2185 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Time-to-first event of the composite endpoint | Approximately 24 months
  Time-to-first event of the composite endpoint consisting of:
  * ESRD (need for chronic dialysis or renal transplantation)
  * Cardiovascular death

SECONDARY OUTCOMES:
Rate of change in estimated glomerular filtration rate (eGFR) over the duration of the study | Approximately 24 months
Time to first hospitalization for heart failure | Approximately 24 months
Time to first event in the composite cardiorenal endpoint | Approximately 24 months
  Time-to-first event in the composite cardiorenal endpoint defined as:
  * Cardiovascular death
  * Non-fatal myocardial infarction
  * Non-fatal stroke
  * Hospitalization for heart failure
Frequency, intensity, and relationship to study drug of adverse events and serious adverse events, as well as clinical and laboratory test abnormalities. | Approximately 24 months

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] de Zeeuw D, Akizawa T, Audhya P, Bakris GL, Chin M, Christ-Schmidt H, Goldsberry A, Houser M, Krauth M, Lambers Heerspink HJ, McMurray JJ, Meyer CJ, Parving HH, Remuzzi G, Toto RD, Vaziri ND, Wanner C, Wittes J, Wrolstad D, Chertow GM; BEACON Trial Investigators. Bardoxolone methyl in type 2 diabetes and stage 4 chronic kidney disease. N Engl J Med. 2013 Dec 26;369(26):2492-503. doi: 10.1056/NEJMoa1306033. Epub 2013 Nov 9. PMID 24206459